CLINICAL TRIAL: NCT03518671
Title: Building a Renewed ImaGe After Head & Neck Cancer Treatment
Acronym: BRIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Evan Graboyes, Associate Professor, Department of Otolaryngology, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 120834
Record Dates: First submitted 2018-04-09; First posted 2018-05-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Body Image Disturbance
Keywords: head and neck cancer; body image disturbance; cognitive behavioral therapy; survivorship
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Cognitive Behavioral Therapy; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT (face to face) (Experimental): Self-limited cognitive behavioral therapy (CBT) delivered via 6 weekly sessions, face-face
  Up to one year after completion of treatment, patients with body image disturbance (BID) as determined by a Body Image Scale (BIS) score > 5 will undergo time-limited CBT consisting of 6 weekly sessions. Each session will be guided by the HNC BID module that we develop but customized to each patient's specific concerns. Each session will last ~60 minutes and be conducted one-one with a psychologist. Patients will complete questionnaires prior to CBT and 1 and 3 months after CBT.
  Interventions: Behavioral: cognitive behavioral therapy, face to face
- CBT (telemedicine) (Experimental): Self-limited cognitive behavioral therapy (CBT) delivered via 6 weekly sessions, via tablet-based telemedicine platform
  Up to one year after completion of treatment, patients with body image disturbance (BID) as determined by a Body Image Scale (BIS) score > 5 will undergo time-limited CBT consisting of 6 weekly sessions. Each session will be guided by the HNC BID module that we develop but customized to each patient's specific concerns. Each session will last ~60 minutes and be conducted one-one with a psychologist. Patients will complete questionnaires prior to CBT and 1 and 3 months after CBT. To overcome the expected travel distance-related barrier to receipt of CBT, patients will receive the intervention via tablet-based telemedicine delivery platform
  Interventions: Behavioral: cognitive behavioral therapy, telemedicine

INTERVENTIONS:
Behavioral: cognitive behavioral therapy, face to face — self-limited cognitive behavioral therapy delivered weekly for 6 weeks via face-face delivery method
  Arms: CBT (face to face)
Behavioral: cognitive behavioral therapy, telemedicine — self-limited cognitive behavioral therapy delivered weekly for 6 weeks via tablet-based telemedicine platform
  Arms: CBT (telemedicine)

SUMMARY:
This study will evaluate whether a time-limited cognitive behavioral therapy (CBT) intervention in the post-treatment time period can address body image disturbance (BID) in patients with surgically-treated head and neck cancer (HNC), thereby improving BID and quality of life (QOL).

DETAILED DESCRIPTION:
The investigators will complete a single-arm, phase II pilot study of time-limited CBT on BID in patients with surgically-treated HNC. Reliable, validated patient-reported outcome (PRO) measures of BID will be collected before, 1 month and 3 months after the CBT intervention to provide preliminary data on the effectiveness of CBT for BID in patients with surgically-treated HNC, addressing this critical knowledge gap. It is expected that time-limited CBT implemented in the post-treatment period will decrease BID and improve QOL in affected patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of squamous cell carcinoma of the upper aerodigestive tract (oral cavity, oropharynx, hypopharynx, larynx) or cutaneous malignancy of the head and neck (e.g. squamous cell, basal cell, melanoma, etc)
* Age > 18
* American Joint Committee on Cancer (AJCC) stages I-IV
* Curative intent therapy with surgery with or without adjuvant therapy
* Body Image Scale (BIS) score > 5 up to 1 year post-treatment

Exclusion Criteria:

* Inability to speak English
* Known distant metastatic disease
* Inability or unwillingness of subject or legal guardian/representative to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Change in Body Image Disturbance | Prior to intervention until 3 months after completion of intervention
  Change in body image disturbance will be measured using Body Image Scale (BIS) scores from before and 3 months after intervention. The BIS has been validated in oncology patients and is the most widely used scale for BID in oncology. It is a 10-item measure that is scored on a 4-point Likert scale; higher scores indicate greater body image dissatisfaction. It addresses the affective, cognitive, and emotional aspects of body image. There are no subscales.

SECONDARY OUTCOMES:
Change in Body Image Investment | Prior to intervention until 3 months after completion of intervention.
  Body image investment (i.e. the importance and influence of appearance) will be measured using the Appearance Schemas Inventory-Revised (ASI-R). This 20-item measure is scored using a 5-point Likert scale with greater scores indicating greater body image investment. There are no subscales.
Change in Body Image Coping Strategies | Prior to intervention until 3 months after completion of intervention
  Change in Body Image Coping strategies will be measured using the Body Image Coping Strategies Inventory (BICSI), a validated measure used to assess cognitive and behavioral responses to manage threats to body image. The subscales are "Appearance Fixing" (10 specific items on the scale), "Avoidance" (8 specific items on the scale), and "Positive Rational Acceptance" (11 items on the scale). Each subscale score is calculated as the mean of the items within that subscale.
Change in Quality of Life | Prior to intervention until 3 months after completion of intervention
  We will employ the European Organisation for Research and Treatment of Cancer (EORTC) QLQ C30/H&N35 module to evaluate quality of life (QOL). The EORTC quality of life questionnaire (QLQ) is an integrated system for assessing the health-related quality of life (QOL) of cancer patients participating in international clinical trials.

OTHER OUTCOMES:
Change in Shame and Stigma | Prior to intervention until 3 months after completion of intervention
  Change in shame and stigma will be measured using the Shame and Stigma Scale, a 20-item, validated tool that measures shame with appearance, stigma, regret, and social/speech concerns in patients with HNC.
Change in Depression and Anxiety | Prior to intervention until 3 months after completion of intervention
  Change in Depression and Anxiety will be measured using Patient-Reported Outcomes Measure Information System (PROMIS), a validated questionnaire developed by the NIH for evaluating health-related quality of life.
Change in Social Roles and Isolation | Prior to intervention until 3 months after completion of intervention
  Social roles and isolation will be assessed by Patient-Reported Outcomes Measure Information System (PROMIS) measures, a validated questionnaire developed by the NIH for evaluating health-related quality of life.
Change in Head and Neck Performance Status and Function | Prior to intervention until 3 months after completion of intervention
  This outcome will be measured by the Performance Status Scale for Head & Neck Cancer, which assesses performance in domains of eating, speech, and diet.
Effectiveness of CBT and Telemedicine Utilization Patterns | One month after completion of study intervention
  We will collect data from patients to understand why they chose face-face CBT versus telemedicine.
Qualitative Assessment of Experience with BID and CBT | One month after completion of study intervention
  To better understand patient experiences with BID not captured in the questionnaires as well as their experiences with CBT, we will perform semi-structured interviews. Participants will be asked to 1) discuss their preferences about the timing, format and content of the CBT sessions 2) describe their program experiences and offer recommendations to improve delivery, and 3) and assess feasibility and acceptability of the intervention. This mixed methods approach will allow for an in-depth exploration of patient experiences, help refine the study intervention, and inform intervention implementation for future studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No